CLINICAL TRIAL: NCT05260658
Title: A Randomized, Double-blind, Placebo-controlled Study of the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Oral Doses of CFTX-1554 in Healthy Subjects, With Comparison of Intake of CFTX-1554 as Liquid Formulation and as Capsule, and After a High-fat Breakfast Versus Fasted
Brief Title: Safety and Tolerability of CFTX-1554 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Confo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CFTX1554-C101; 2021-006368-26 (EudraCT Number)
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: CFTX-1554 Single Ascending Dose (SAD) (Experimental): Up to 7 dose levels with CFTX-1554 administered as oral liquid formulation under fasted conditions (at 1 single dose level only, drug intake under fed conditions, and as capsule under fasted conditions and under fed conditions, will be assessed)
  Interventions: Drug: CFTX-1554
- Part A placebo (Placebo Comparator): Single placebo administration in study Part A
  Interventions: Drug: Placebo
- Part B: CFTX-1554 Multiple Ascending Dose (MAD) (Experimental): Up to 4 dose levels with CFTX-1554 in Part B. Doses and dosing frequency will be decided based on the results of study Part A.
  Interventions: Drug: CFTX-1554
- Part B placebo (Placebo Comparator): Multiple placebo administration in study Part B
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CFTX-1554 — CFTX-1554 is a new chemical entity that binds to the angiotensin II type 2 receptor (AT2R).
  Arms: Part A: CFTX-1554 Single Ascending Dose (SAD); Part B: CFTX-1554 Multiple Ascending Dose (MAD)
Drug: Placebo — CFTX-1554 matching placebo
  Arms: Part A placebo; Part B placebo

SUMMARY:
The study will consist of 2 parts, i.e. a single ascending dose part with integrated food effect assessment and assessment of relative bioavailability (Part A), and a multiple ascending dose part (Part B).

Part A will have a randomized, double-blind, placebo-controlled design. Subjects will receive single ascending doses of CFTX-1554 or placebo (as liquid formulation under fasted condition) in 7 subsequent cohorts. Drug intake under fed conditions, and as capsule under fasted conditions and under fed conditions (Periods 2 to 4), compared to liquid formulation under fasted conditions (Period 1) (1 single dose level only) will be assessed.

Part B will have a randomized, double-blind, placebo-controlled design, assessing multiple ascending oral doses of CFTX-1554 or placebo in 4 subsequent cohorts.

ELIGIBILITY:
INCLUSION CRITERIA:

* Body mass index 18.0 to 30.0 kg/m2
* Females may be of childbearing potential but not pregnant or lactating, or of nonchildbearing potential; all females will be required to have a negative serum pregnancy test conducted at screening, (each) admission, and follow-up.
* Female subjects of childbearing potential who have a fertile male sexual partner must agree to use adequate contraception from at least 4 weeks prior to first administration of study drug until 90 days after the follow up visit.
* Male subjects, if not surgically sterilized, must agree to use adequate contraception and not donate sperm from first admission to the clinical research center until 90 days after the follow-up visit.
* All prescribed medication must have been stopped at least 30 days prior to first admission to the clinical research center.
* All over-the-counter medication, vitamin preparations and other food supplements, or herbal medications must have been stopped at least 14 days prior to first admission to the clinical research center.
* Ability and willingness to abstain from alcohol from 48 hours before screening and first admission to the clinical research center.
* Ability and willingness to abstain from methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, energy drinks) and grapefruit (juice) from 48 hours before first admission to the clinical research center.
* Good physical and mental health on the basis of medical history, physical examination, clinical laboratory, ECG, and vital signs, as judged by the Investigator.
* Willing and able to sign the Informed Consent Form.

EXCLUSION CRITERIA:

* Previous participation in the current study
* History of relevant drug and/or food allergies
* Allergy or hypersensitivity to active ingredient or excipients of the study drug
* Using nicotine-containing products within 60 days prior to the first study drug administration
* History of alcohol abuse or drug addiction (including soft drugs like cannabis products) within 1 year before screening
* Positive drug and alcohol screen in urine (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants, nicotine metabolites [cotinine], and alcohol) at screening or at one of the admissions to the clinical research center
* Average intake of >24 units of alcohol/week
* Positive screen for hepatitis B surface antigen, hepatitis C virus antibodies, or human immunodeficiency virus 1 and 2 antibodies
* Participation in a drug study within 30 days prior to the first study drug administration in the current study (counting from the follow-up visit to the screening visit). Participation in ≥4 other drug studies in the 12 months before the first study drug administration in the current study
* Donation or loss of >450 mL of blood within 60 days pribefore the first study drug administration. Donation or loss of >1.5 L of blood in male subjects) or >1.0 L of blood in female subjects in the 10 months before the first study drug administration in the current study.
* Significant and/or acute illness within 5 days before the first study drug administration that may impact safety assessments, in the opinion of the Investigator.
* Unwillingness to consume the Food and Drug Administration (FDA) breakfast or intolerance to any of the ingredients of the FDA breakfast (Cohort A5 only)
* Vaccination against SARS-CoV-2 planned between 2 weeks before first admission and follow-up.
* Positive nasopharyngeal PCR test for SARS-CoV-2 on Day -1, or any known contact with a person who tested positive for SARS-CoV-2 or with a COVID 19 patient within 2 weeks before admission.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | Day -1 through Day 13 (Single Ascending Dose study part) or Day 26 (Multiple Ascending Dose study part)
  Number of Participants With Adverse Events Following Oral Administration of CFTX-1554 in SAD (Part A) and MAD (Part B)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Vicini, PhD, Study Chair — Confo Therapeutics
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No